CLINICAL TRIAL: NCT03750448
Title: Does Rehabilitation After Total Hip and Knee Arthroplasty Work: A Pragmatic, Randomised, Controlled, Superiority Trial (The DRAW1 Trial)
Brief Title: Does Rehabilitation After Total Hip and Knee Arthroplasty Work
Acronym: DRAW1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bornholms Regionskommune (Other Government)
Responsible Party: Principal Investigator, Troels Mark Christensen, Principal investigator, Bornholms Regionskommune
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56929866
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip; Telerehabilitation; Rehabilitation
Keywords: Total knee arthroplasty; Total hip arthroplasty; Randomized controlled trial; No intervention; Telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Telerehabilitation.
  No intervention.
  Unsupervised rehabilitation.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: A physiotherapist will assess the outcomes at baseline after which the patients are randomized. The same physiotherapist will then deliver the allocated intervention and no longer assess outcomes for this patient. A different physiotherapist, who is blinded to treatment allocation, will assess outcomes at the follow-up visits in this patient. At all follow-up visits, patients will be asked not to disclose any information regarding group allocation, and the physiotherapists will be instructed not to ask questions regarding group allocation.
  The patients are blinded to the trial hypothesis in order to prevent ascertainment bias. The principal investigator is not an outcome assessor and will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation (Active Comparator): Patients randomized to this group will receive interactive virtual rehabilitation using a mobile app. The telerehabilitation is based on sensor technology, developed by ICURA. This technology consists of motion sensors that can measure and analyse the quantity and quality of the exercises, and a mobile application that can guide the patient with visual response. A unique feature of ICURA trainer allows the physiotherapist to remotely supervise the individual patients exercise adherence and progress. This technology has already been successfully implemented in several different rehabilitation facilities across Denmark, and, hence, reflects current clinical practice.
  Interventions: Other: Telerehabilitation
- No intervention (Active Comparator): This group of randomised patients will not be given any physical rehabilitation intervention. This means no physical activity or exercise designed and prescribed for restoring normal function or reducing pain cause by disease, injury or surgery. The no intervention group will be encouraged to stay active and continue life as usual, gradually returning to their activities of daily living when they feel ready for it.
  Interventions: Other: No intervention
- Unsupervised rehabilitation (Active Comparator): This group will be instructed in similar exercises as patients allocated to telerehabilitation. However, this group will receive a written exercise-program with instructions to perform these exercises at home. The home-based exercise program will be created using exercise templates from Exorlive. Using a link provided in the exercise-program, the patients will be able to see short instruction-videos of the individual exercises.
  Interventions: Other: Unsupervised rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The telerehabilitation intervention is based on sensor technology, developed by ICURA. The technology consists of motion sensors that can measure and analyse the quantity and quality of the exercises, and a mobile application that can guide the patients with visual response. A unique feature of ICURA trainer allows the physiotherapist to remotely supervise the individual patients exercise adherence and progress. The patients will receive a suitcase with five sensors (to be placed bilaterally on lower legs, thighs and one around the waist), a smartphone to record the exercises and a charging station free of charge during the 6-week intervention. At the end of the intervention the material will be returned at the first follow-up (t1). For more information please visit https://icura.dk.
  Arms: Telerehabilitation
Other: No intervention — Patients allocated to the no intervention group will receive encouragement to stay active and be encouraged to gradually return to activities of daily living. This will be the only exercise-encouragement given to the no-intervention group.
  Arms: No intervention
Other: Unsupervised rehabilitation — The unsupervised rehabilitation group will receive a written exercise program in order to perform daily exercises at home. The exercise program will be made using Exorlive (for more information about Exorlive please visit https://www.exorlive.com). In addition to the written program, patients will able to use a link provided to see small video-instructions on the internet of each exercise on the program. No feedback or supplementary instructions will be given after the initial face-to-face appointment.
  Arms: Unsupervised rehabilitation

SUMMARY:
Background: Total hip- and knee arthroplasty (THA and TKA) is recommended for relieving pain and restoring function for end-stage osteoarthritis, when non-surgical treatment has failed to relieve symptoms. Following THA and TKA post-discharge physical rehabilitation is common practice, but vary significantly regarding content, duration, intensity and mode of delivery. Recent systematic reviews have found home-based rehabilitation to be as good as outpatient rehabilitation in terms of pain and physical function. Additionally, no long-term benefits seem to persist compared to minimal or no intervention following THA or TKA; questioning the true effectiveness of postoperative rehabilitation. However, a true "no intervention" (e.g. no prescribed exercises) has never been investigated following total THA or TKA. The purpose of this present trial is to compare the effectiveness of telerehabilitation, unsupervised rehabilitation and no rehabilitation to enhance recovery following THA and TKA.

Methods: This pragmatic, randomised controlled trial will include 168 patients following discharge after THA or TKA. Patients will be randomized into one of the three 6-week interventions: telerehabilitation, unsupervised rehabilitation or no intervention. The trial is designed as a superiority trial to test the hypothesis that rehabilitation (telerehabilitation and unsupervised rehabilitation) is superior to no rehabilitation. The primary outcome will be the difference between intervention groups in terms of the mean score of the Hip disability and Osteoarthritis Outcome Score (HOOS)/ the Knee injury and Osteoarthritis Outcome Score (KOOS)-subscale: function of daily living at first follow-up (end of the 6-week intervention). Additional follow-up are scheduled at 3 and 12 months. Outcome assessors and data analysts are blinded to group allocation.

Discussion: As the number of THA and TKA procedures are expected to increase, the need to find effective postoperative rehabilitation strategies are warranted. Knowledge on the effectiveness of the three investigated rehabilitation strategies will help guide the future direction of post-discharge rehabilitation following THA and TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients having had primary, unilateral THA or TKA due to osteoarthritis.
* Patients being referred to receive postoperative rehabilitation at our institution.
* Patients being able to speak, read and understand Danish language.
* Patients aged ≥ 18 years.

Exclusion Criteria:

* Patients not able to comply with exercise instructions.
* Patients who are discharged to a nursing-home facility or receiving in-home rehabilitation by home care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
For THA's: Hip disability and Osteoarthritis Outcome Score (HOOS) subscale: function in daily living (ADL). | Difference between groups at first follow up (6 weeks)
  This subscale consists of 17 questions related to the patient's function in activities of daily living such as "descending stairs", "standing" and "getting in/out of car". The subscale is scored by the degree of difficulty the patient experiences in the last week on a 5-point Likert scale (none, mild, moderate, severe, and extreme), and calculated to a score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). The total questionnaire takes about 10 minutes to complete. At least 50% of the questionnaire items are required to be answered to permit calculation of a mean score.
For TKA's: Knee injury and Osteoarthritis Outcome Score (KOOS) subscale: function in daily living (ADL). | Difference between groups at first follow up (6 weeks)
  This subscale consists of 17 questions related to the patient's function in activities of daily living such as "descending stairs", "standing" and "getting in/out of car". The subscale is scored by the degree of difficulty the patient experiences in the last week on a 5-point Likert scale (none, mild, moderate, severe, and extreme), and calculated to a score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). The total questionnaire takes about 10 minutes to complete. At least 50% of the questionnaire items are required to be answered to permit calculation of a mean score.

SECONDARY OUTCOMES:
For THA's: Hip disability and Osteoarthritis Outcome Score (HOOS) subscale: function in daily living (ADL). | Difference between groups at 3 and 12 months follow up.
  This subscale consists of 17 questions related to the patient's function in activities of daily living such as "descending stairs", "standing" and "getting in/out of car". The subscale is scored by the degree of difficulty the patient experiences in the last week on a 5-point Likert scale (none, mild, moderate, severe, and extreme), and calculated to a score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). The total questionnaire takes about 10 minutes to complete. At least 50% of the questionnaire items are required to be answered to permit calculation of a mean score.
For TKA's: HKnee injury and Osteoarthritis Outcome Score (KOOS) subscale: function in daily living (ADL). | Difference between groups at 3 and 12 months follow up.
  This subscale consists of 17 questions related to the patient's function in activities of daily living such as "descending stairs", "standing" and "getting in/out of car". The subscale is scored by the degree of difficulty the patient experiences in the last week on a 5-point Likert scale (none, mild, moderate, severe, and extreme), and calculated to a score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). The total questionnaire takes about 10 minutes to complete. At least 50% of the questionnaire items are required to be answered to permit calculation of a mean score.
For THA's: Hip disability and Osteoarthritis Outcome Score (HOOS) subscale: symptoms, pain and hip- or knee related quality of life. | Baseline, follow up at 6 weeks, 3 and 12 months.
  These subscales are scored by the degree of difficulty the patient has experienced in the last week on a 5-point Likert scale. Each subscale provides a score, which can be calculated to a total score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). At least 50% of the questionnaire items in each subscale are required to be answered to permit calculation of a mean score.
For TKA's: Knee injury and Osteoarthritis Outcome Score (KOOS) subscales: symptoms, pain and hip- or knee related quality of life. | Baseline, follow up at 6 weeks, 3 and 12 months.
  These subscales are scored by the degree of difficulty the patient has experienced in the last week on a 5-point Likert scale. Each subscale provides a score, which can be calculated to a total score ranging from 0 (worst/extreme difficulties) to 100 (best/ no problems). At least 50% of the questionnaire items in each subscale are required to be answered to permit calculation of a mean score.
Patient global assessment. | Baseline, follow up at 6 weeks, 3 and 12 months.
  At baseline the patient's perception of his or her overall functional ability will be assessed using a single numeric rating scale, as recommended by OARSI. The patient will be asked a single question: "How would you rate your current level of function during your usual activities of daily living?" During follow-up assessment patients will be asked the same question as at baseline. Their answer will be rated on a 0-100 visual rating scale with end-points anchored as "Inability to perform any daily activities" (0) and "No problem with any daily activity" (100)
30-s chair stand test. | Baseline, follow up at 6 weeks, 3 and 12 months.
  Performance-based assessment will be performed using the 30-s chair-stand test, which represent the sit-to-stand activity. The test counts the number of sit-to-stand repetitions the patient can perform in 30 seconds. The straight-back chairs used for testing during all outcome assessments will be of the same model, same height (approximately 43 cm), and will be placed against a wall. Any other adaptations (i.e. the use of armrests or assistive devices) will be reported. To assure understanding, two slow-paced repetitions will be practiced before the test initiates. The 30-s chair stand test has proven good reliability to measure functional performance following THA and TKA.
40 meters walking test. | Baseline, follow up at 6 weeks, 3 and 12 months.
  This performance-based assessment measures short distance walking activity. The patient will be instructed to walk as quickly as safely as possible to a mark 10 meters away, return and repeat for a total distance of 40 meters. Each walk of 10 meters (excluding the turn time) is recorded and expressed as speed m/s by dividing distance by time in seconds. A practice walk up and back will be performed to assure understanding. Any assistive devices used will be recorded.
Use of analgesics. | Baseline, follow up at 6 weeks, 3 and 12 months.
  The use of analgesics will recorded at baseline and at all follow-up assessments, using a nominal scale (yes/no) regarding the daily consumption of opioids, non-steroid-anti inflammatorily drug (NSAID) and paracetamol. If the patient were not aware of his or hers use of analgesics, a medical record will obtained to assess the use of analgesics.
Type of walking assistant devices. | Baseline, follow up at 6 weeks, 3 and 12 months.
  The type (e.g. elbow crutches, walker) will be recorded. The need for walking assistant devices will be assessed by what the patient use during normal activities of daily living.
Patient satisfaction.: 4-Likert ordinal scale | Follow up at 6 weeks.
  Patients will be asked to answer four questions to indicate their level of satisfaction. The answers will be based on a 4-Likert ordinal scale with the categories: very satisfied (100 points), somewhat satisfied (75 points), somewhat dissatisfied (50 points), and very dissatisfied (25 points). The score is the unweighted mean of the combined scores. The four questions are: "How satisfied are you with the results of your surgery and rehabilitation?", "How satisfied are you with your surgery and rehabilitation for improving your pain?", "How satisfied are you with the results of your surgery and rehabilitation for improving your ability to do home or yard work?" and "How satisfied are you with the results of surgery and rehabilitation for improving your ability to do recreational activities?". The questions are modified from the Self-Administered Patient Satisfaction Scale for Primary Hip and Knee Arthroplasty.
Time usage (care provider). | Baseline, follow up at 6 weeks, 3 and 12 months.
  Analysis of the economical resources required for each of the three rehabilitation strategies. The principal investigator intend to use this data in a later cost-analysis.
Number of adverse events. | Baseline, follow up at 6 weeks, 3 and 12 months.
  Number and nature of adverse events during enrolment of the trial will be recorded, regardless of the relation to the trial.

OTHER OUTCOMES:
For telerehabilitation group: Exercise adherence | Follow up at 6 weeks.
  Exercise adherence will be measured as a percentage (0-100), where 0 % indicates total non-adherence and 100 % indicates total adherence to the exercise prescription. Exercise adherence is objectively recorded in the telerehabilitation group and can be extracted from the device used by the patients.
Exercise adherence. | Follow up at 6 weeks.
  Exercise adherence will be measured as a self-reported percentage (0-100), where 0 % indicates total non-adherence and 100 % indicates total adherence to the exercise prescription. The patients will be asked: "What percentage of the prescribed 42 exercise sessions (one exercise session per day for 6 weeks; corresponding to 100 %) have you completed the past 6 weeks?". The scale will be illustrated with a 0-100mm visual rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Q. Bandholm, Phd., Study Director — Physical Medicine and Rehabilitation Research-Copenhagen (PMR-C); Department of Physical and Occupational Therapy; Clinical Research Centre; Department of Orthopaedic Surgery, Hvidovre Hospital, University of Copenhagen, Hvidovre Denmark
Locations (3):
- Denmark (3):
  - NMC Rehabilitation, Nexø, Bornholm
  - Lunden Rehabilitation, Rønne, Bornholm
  - Sønderbo Rehabilitation, Rønne, Bornholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mark-Christensen T, Thorborg K, Kallemose T, Bandholm T. Clinical benefit of physical rehabilitation after total hip and knee arthroplasty: A pragmatic, randomized, controlled trial (The DRAW1 trial). Osteoarthr Cartil Open. 2024 Oct 16;6(4):100530. doi: 10.1016/j.ocarto.2024.100530. eCollection 2024 Dec. PMID 39507936
- [Derived] Mark-Christensen T, Thorborg K, Kallemose T, Bandholm T. Physical rehabilitation versus no physical rehabilitation after total hip and knee arthroplasties: Protocol for a pragmatic, randomized, controlled, superiority trial (The DRAW1 trial). F1000Res. 2021 Feb 25;10:146. doi: 10.12688/f1000research.50814.2. eCollection 2021. PMID 34316356